CLINICAL TRIAL: NCT03361579
Title: Pain Response to Open Label Placebo in Induced Acute Pain in Healthy Male Adults - A Randomized Single Blinded Clinical Trail
Brief Title: Pain Response to Open Label Placebo in Induced Acute Pain in Healthy Male Adults
Acronym: POLAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-01690
Record Dates: First submitted 2017-11-17; First posted 2017-12-05 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Acute Pain
Keywords: Placebo
MeSH Terms: conditions — Acute Pain | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: investigator blinded, cross over design
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator is blinded about the source of education a participant recieved prior to Placebo application. Investigator is blinded about during which Intervention the Placebo is applicated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo education group (Other): Prior to the intervention during the Placebo is given, the volunteer receives a detailed information about the effect and the strength of an open-label placebo. This education is performed via a slide show and a news report video. The important terms for Placebo analgesia: positive expectations, conditioning, communication are discussed
  Interventions: Other: Education
- Placebo non education group (Other): No detailed Information about open-label placebo prior to the intervention. The volunteer is told about the possible strength of the Placebo effect on pain directly before the application.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — c.p. intervention description

SUMMARY:
Open Label Placebo application has been shown to be effective in treatment of chronic pain (low back pain) and disease like the irritable bowel Syndrome. Data about effects on acute pain are spare.

The study investigates the effect of an open-label Placebo (substance without a medical active component) application on acute pain, evoked via a artificial pain model in healthy male volunteers. 32 healthy male volunteers are recruited.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers (American Society of Anaesthesiologist's Class I or II)
* Body mass index between 18 and 25kg/m2
* Able to understand the study and the NRS scale
* Able to give informed consent

Exclusion Criteria:

* Recreational drug abuse
* Regularly taking medication potentially interfere with pain sensation (analgesics, antihistamines and calcium and potassium channel blockers)
* Neuropathy
* Chronic pain
* Neuromuscular or psychiatric disease
* Known or suspected kidney or liver disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Pain response measured by the Area under the Pain Curve (AUPC) | 30 minutes after baseline until 100 minutes after baseline
  Pain response measured by creating the Area under the Pain Curve (AUPC), using the numeric rating scale (NRS) from minute 30 to 100 during constant induced pain with electrical current at the forearm of the participant. Measuring of pain every 10 minutes from minute 30 to 100 (Minute 30,40,50,60,70,80,90, 100) in an experimental setting. Main comparison: The effect of open label placebo v.s. no treatment intervention

SECONDARY OUTCOMES:
Differences in pain response measured by the AUPC due to education | 30 minutes after baseline until 100 minutes after baseline
  The pain response measured by the AUPC in participants received a detailed education about open label Placebo compared to those who received a short education direct prior to placebo administration.
hyperalgesia | 100min
  Hyperalgesia will be measured analogously to the NRS
Saliva cortisol concentration in μg/dL | baseline until 100 min after baseline
  Saliva concentration of cortisol, will be measured 4 times: at baseline, 30, 60 and 100 minutes during pain induction
allodynia | 100minutes
  allodynia will be measured analogously to the NRS

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Ruppen, PD, Study Director — Dep. Anesthesiology University Hospital Basel
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT03361579/Prot_SAP_000.pdf